CLINICAL TRIAL: NCT02200081
Title: Randomized Clinical Study of Maintenance Therapy With Immunomodulator MGN1703 in Patients With Extensive Disease Small Cell Lung Cancer After Platinum-Based First-Line Therapy
Brief Title: Randomized Study of Maintenance Therapy With MGN1703 in Patients With SCLC
Acronym: IMPULSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mologen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGN1703-C03
Record Dates: First submitted 2014-01-09; First posted 2014-07-25 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Small Cell Lung Cancer
Keywords: Extensive disease; After first line therapy; Immuno therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — MGN1703; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MGN1703 (Experimental): MGN1703, solution in Dulbecco's Phosphate-Buffered Saline (DPBS), 2 mL of 60 mg/4 mL (15 mg/mL), administered SC at 2 application sites twice weekly
  Interventions: Drug: MGN1703
- Standard of care (Other): Continous first line therapy
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: MGN1703
  Other Names: dSLIM
  Arms: MGN1703
Other: Standard of care — Usual Standard of Care according to local investigators practise, e.g. Treatment break continous treatment and other
  Arms: Standard of care

SUMMARY:
Evaluation of efficacy and safety of MGN1703 administered twice weekly subcutaneously (SC) as maintenance treatment in patients with extensive disease small cell lung cancer (SCLC) who achieved at least a partial response (PR) following platinum-based first-line therapy.

ELIGIBILITY:
1. Male and female patients with extensive disease SCLC ≥ 18 years of age receiving first line treatment;
2. Histology of SCLC or mixed histology of SCLC if SCLC histology is at least 80%;
3. Completion of 4 cycles of first-line therapy with a platinum-based regimen and no other prior chemotherapy;
4. Documented evidence of tumor response as assessed by investigators after the first 2 cycles of platinum-based chemotherapy followed by a confirmed PR or CR at the end of fourth cycle by CT or MRI scan;
5. Brain metastases are allowed only after cranial irradiation, if not requiring continuous treatment with steroids or anticonvulsants;
6. ECOG performance status 0 or 1;
7. Adequate organ function with total bilirubin, lactate dehydrogenase [LDH], alkaline phosphatase [AP], gamma glutamyltransferase [GGT], albumin, creatinine, urea, electrolytes, and coagulation parameters ≤ 1.5 × upper limit of normal (ULN), and with aspartate aminotransferase [AST] and ALT ≤ 2.5 × ULN in the absence of liver metastases or ≤ 5.0 × ULN in the presence of liver metastases;
8. Adequate hematological parameters: absolute neutrophil count ≥ 1.5 × 109/L; platelet count ≥ 100 × 109/L; leukocyte count ≥ 3.0 × 109/L; lymphocytes ≥ 1.0 × 109/L; hemoglobin ≥ 9.0 g/dL or 5.59 mmol/L;
9. Patients with reproductive potential agree to use effective contraceptive measures throughout the study;
10. Negative pregnancy test in women of childbearing potential;
11. Signed informed consent form (ICF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 24 months
  The primary efficacy endpoint is the OS which is defined as the time interval starting with the randomization and lasting until death (=event) or until the date of last information available from the patient.

SECONDARY OUTCOMES:
OS1 | 24 months
  The secondary efficacy endpoint OS1 is defined as the time interval starting at the first cycle of induction therapy and lasting until death (=event) or until the date of last information available from the patient.
  OS1 will be estimated by Kaplan-Meier estimates. The comparison between the treatment groups will be performed using the log-rank test with a significance level of α = 2.5% for the 1-sided test. The OS1 will be presented as Kaplan-Meier figures also.

OTHER OUTCOMES:
Progression-free survival (PFS) PFS from the start of the first cycle of induction therapy (PFS1) ass | 24 months
  Progression-free survival is the time after randomization to either disease progression (PD), measured using RECIST 1.1 and irRC criteria and confirmed via centralized review or death

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Surmont, MD, Principal Investigator — University Hospital Ghent, Belgium 9000; Georg Pall, MD, Principal Investigator — Medizinische Universität Innsbruck, Innere Medizin, Hämatologie und Onkologie
Locations (4):
- Medizinische Universitaet Innsbruck, Innsbruck, Austria
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Thoraxklinik Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg, Germany
- Hospital Universitario Fundación Jiménez Díaz, Madrid, Spain

REFERENCES:
- [Result] Thomas M, Ponce-Aix S, Navarro A, Riera-Knorrenschild J, Schmidt M, Wiegert E, Kapp K, Wittig B, Mauri C, Domine Gomez M, Kollmeier J, Sadjadian P, Frohling KP, Huber RM, Wolf M; IMPULSE study team. Immunotherapeutic maintenance treatment with toll-like receptor 9 agonist lefitolimod in patients with extensive-stage small-cell lung cancer: results from the exploratory, controlled, randomized, international phase II IMPULSE study. Ann Oncol. 2018 Oct 1;29(10):2076-2084. doi: 10.1093/annonc/mdy326. PMID 30137193